CLINICAL TRIAL: NCT00581061
Title: Vesicare™ (Solifenacin) in the Treatment of Urinary Incontinence After Radical Prostatectomy
Brief Title: Study to Determine Effects of Vesicare on Return to Continence Post- Radical Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study subjects were not compliant with study protocols.
Sponsor: University of California, Irvine (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Thomas Ahlering, MD, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-5720
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2010-09-30 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Incontinence
Keywords: Incontinence; Robotic Prostatectomy
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vesicare Treatment (Experimental)
  Interventions: Drug: Vesicare

INTERVENTIONS:
Drug: Vesicare — Vesicare will be taken daily for one or three months, depending on symptoms of subject.
  Other Names: Solifenacin

SUMMARY:
Prostate cancer is the most common non-cutaneous malignancy in men and is the 2nd leading cause of death from cancer in men. Radical prostatectomy is one of the treatment options available for organ-confined disease. Over 100,000 radical prostatectomies cases (total removal of the cancerous prostate by surgery) are performed in the United States yearly. Unfortunately nearly all of the men undergoing surgery report diminished Quality of Life (QOL) scores due in part due to a postoperative incontinence which may require the use of multiple urinary pads per day. Many of these men also report debilitating irritative voiding symptoms of urinary urgency and frequency, and have overall decreased urinary satisfaction scores. Abatement of these symptoms can take up to one year in men, and in 5-20% of patients symptoms may persist for longer periods.

Our recent published findings suggest that instability in the bladder muscle is likely an underlying etiology in postoperative urinary incontinence. This 'Detrusor Muscle' instability results in excess contractions of the urinary bladder ('urgency to urinate'), and can result in the feeling of needing to urinate more frequently. Consistent with this hypothesis of detrusor muscle instability, men with postoperative dribbling had more complaints with urgency, frequency and bother scores when queried with validated questionnaires. We suspect that a transient bladder muscle contraction may overcome the urinary sphincter valve resistance and result in the patient's dribbling of urine.

By treating the bladder muscle instability, we expect improved postoperative continence and improved quality of life in patients after undergoing surgery for total removal of a cancerous prostate. This pilot study will assess the statistical requirements for the number of subjects needed for a fully 'powered' randomized prospective study to fully evaluate whether medications such as solifenacin significantly improve patients' quality of urinary life and improve postoperative urinary incontinence after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with prostate cancer undergoing robotic radical prostatectomy
* Incontinence
* Obesity
* Large prostate weight
* Mild and severe AUA symptom scores
* Urinary Bother

Exclusion Criteria:

* Contra-indication to Solifenacin
* Narrow angle glaucoma
* Hepatic impairment
* Renal impairment
* CYP3A4 inhibitors (e.g. Ketoconazole)
* Gastric Retention (delayed or slow emptying of the stomach)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ahlering, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vesicare: Number of subjects that were in compliance with the study protocol and took medication for at least one month.
Period: Overall Study
Arm/Group | Vesicare
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vesicare
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Continence
Description: Time in days to achieve pad free urinary continence
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Vesicare: Number of days it takes for subjects to achieve pad free urinary continence
Arm/Group | Vesicare
Number analyzed (Participants) | 10
days | 50 (2.5)

2. Secondary Outcome: Compliance
Description: Number of subjects that were in compliance with the study protocol and took medication for at least one month.
Time Frame: 3 months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Vesicare
Number analyzed (Participants) | 13
participants | 10

3. Secondary Outcome: Side Effects
Description: Number of people who experienced side effects while taking Vesicare, per study protocol.
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Vesicare: Number of people who experienced side effects while taking Vesicare, per study protocol. These are known side effects indicated on the drug label that occur to subjects on this medication.
Arm/Group | Vesicare
Number analyzed (Participants) | 10
participants
  Constipation | 2
  Fatigue | 1
  Heartburn | 1
  Dry Hands | 1
  Dry Mouth | 2

ADVERSE EVENTS:
Arm/Group | Vesicare
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vesicare (N=13)
Constipation (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Dry Hands (Skin and subcutaneous tissue disorders) | 1
Dry Mouth (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less